CLINICAL TRIAL: NCT01487330
Title: First In Human Experience and Assessment of the 23mm SJM Transcatheter Aortic Valve Implant and the SJM TAVI Transfemoral Delivery System (SJM TAVI FIH)
Brief Title: First in Human Experience of the St. Jude Medical TAVI Valve and Delivery System
Acronym: SJM TAVI FIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1103
Record Dates: First submitted 2011-08-01; First posted 2011-12-07 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Symptomatic Aortic Stenosis
Keywords: aortic stenosis; aortic valve stenosis; valvular heart disease; aortic valve replacement; transcatheter aortic valve implantation; TAVI; TAVR
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects receiving TAVI valve (Experimental)
  Interventions: Device: Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation (TAVI) — Placement of the SJM TAVI aortic valve with a transfemoral delivery system.

SUMMARY:
The purpose of this first-in-human study is to assess the technical feasibility, deployment characteristics, and safety of the 23mm SJM Transfemoral Transcatheter Heart Valve and delivery system in subjects with severe symptomatic aortic stenosis (AS).

This is a single center, prospective, non-randomized, first-in-human investigational study without concurrent or matched controls.

DETAILED DESCRIPTION:
Data will be collected at baseline, procedure, discharge (date of hospital discharge or 7 days post-implant, whichever occurs first), 30 days post implant, 3 months post implant, 6 months post implant, and 12 months post implant.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent for participation prior to procedure.
2. Legal age in host country.
3. Aortic annulus 19-21mm diameter
4. Senile degenerative aortic stenosis with derived mean gradient >40mmHg or jet velocity greater than 4.0 m/s or an initial valve area of <1.0 cm2 (or aortic valve area index ≤ 0.6 cm2/m2)
5. NYHA Functional Classification of II or greater.
6. Predicted operative mortality or serious, irreversible morbidity risk is <50% at 30 days.
7. Suitable peripheral vessels and aorta to allow for access of the 18 French delivery system.

Exclusion Criteria:

1. History of a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months (≤180 days) of index procedure.
2. Carotid artery disease requiring intervention.
3. Myocardial infarction (MI) within 6 months (≤180 days) of the index procedure.
4. Native aortic valve that is congenitally unicuspid, bicuspid, quadricuspid or non-calcified as seen by echocardiography.
5. Mitral or tricuspid valvular regurgitation (grade II) or moderate to severe mitral stenosis.
6. Aortic root angulation >70 degrees (horizontal aorta).
7. Pre-existing prosthetic valve or prosthetic ring in any position. LVEF < 20%.
8. Untreated coronary artery disease (CAD) requiring revascularization.
9. Severe basal septal hypertrophy.
10. Percutaneous interventional or other invasive cardiac or peripheral procedure ≤ 14 days or history of previous endocarditis.
11. Uncontrolled atrial fibrillation (AF) or is in chronic AF without long term oral anticoagulation.
12. Evidence of intracardiac mass, thrombus, or vegetation.
13. Hemodynamic instability
14. Significant pulmonary disease.
15. Nonreactive pulmonary hypertension.
16. Chronic steroid use.
17. Hypersensitivity or contraindication to anticoagulant or antiplatelet medication.
18. Renal insufficiency as evidenced by a serum creatinine > 3.0 or end-stage renal disease requiring chronic dialysis.
19. Morbid obesity defined as BMI ≥ 35.
20. Subject's iliac arteries have severe calcification, tortuosity, diameter <6mm, or subject has had an aorto-femoral bypass.
21. Ongoing infection or sepsis.
22. Blood dyscrasias
23. Significant aortic disease.
24. Pre-existing endovascular stent graft in the supra- or infrarenal aorta or pre-existing stent grafts in the ileo-femoral arteries.
25. Active peptic ulcer or has had gastrointestinal (GI) bleeding within the past 3 months (≤ 90 days) prior to the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Assessment of Technical Feasibility and Device Deployment Characteristics | At time of procedure
  Evaluate the technical feasibility and device deployment characteristics (observed at procedure) by:
  1. The ability for the valve to be deployed at the desired location
  2. The ability to complete the full procedure
  3. Quantification of the time from delivery system entry to a fully deployed and functional valve

SECONDARY OUTCOMES:
Quantification of SAEs Reported (Device Related or Procedure Related) | Through 12 months post implantation
  Evaluate the safety of the 23mm SJM Transcatheter Aortic Heart Valve and transfemoral delivery system by:
  1. Summarizing the SAEs observed at procedure that are device or procedure related
  2. Summarizing the SAEs observed during the study

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Manoharan, MD, Principal Investigator — Royal Victoria Hospital, Belfast
Locations (1):
- Royal Victoria Hospital, Belfast, United Kingdom